CLINICAL TRIAL: NCT01382823
Title: Laser Cataract Surgery With the Femtosecond Laser Technology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Melissa Earl, CRO
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMTO 2010
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Femtosecond Laser (Experimental)
  Interventions: Procedure: Femtosecond Laser

INTERVENTIONS:
Procedure: Femtosecond Laser — Using the Femtosecond Laser to make a clear corneal incision.

SUMMARY:
The purpose of this study is to prove the efficacy and safety of the Femtosecond laser to create a clear corneal incision during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have a cataract for which phacoemulsification extraction and posterior IOL implantation has been planned in at least one eye.
* Study participants should be capable of achieving better than 20/30 Snellen best corrected distance vision after cataract extraction and IOL implantation.
* The surgeon may use the Mento Potential Acuity Meter (PAM)laser interferometer, McIntyre Pinhole, or his/her judgement to estimate the patient's potential acuity.

Exclusion Criteria:

* Concurrent participation or participation in the last 30 days in other clinical trials.
* Known steroid IOP responder.
* Taking medications that may affect vision, IOP, or ease of cataract surgery (e.g. Flomax, Glaucoma medications, etc.).
* Acute or chronic disease or illness that would increase risk or confound study results(e.g. uncontrolled diabetes mellitus, immunocompromised, etc.).
* Uncontrolled systemic or ocular disease.
* Corneal abnormalities (e.g. stromal, epithelial, or endothelial dystrophies)
* Pseudoexfoliation.
* Ocular hypertension (>or =20hg) or glaucomatous changes in the optic nerve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | three month
  Measure the fluid pressure inside the eye.
Uncorrected and Best corrected Visual Acuity | three month
  Vision obtained with the best possible lens correction (Best corrected). Vision obtained without the use of glasses or contact lenses (Uncorrected).

CONTACTS AND LOCATIONS:
Overall Officials: James Loden, MD, Principal Investigator — Loden Vision Centers
Locations (1):
- Loden Vision Centers, Goodlettsville, Tennessee, United States